CLINICAL TRIAL: NCT06356662
Title: Efficacy and Safety of Tenofovir Disoproxil Fumarate in the Treatment of Parkinson's Disease
Brief Title: Tenofovir Disoproxil Fumarate in the Treatment of Parkinson's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2023-198
Record Dates: First submitted 2024-03-27; First posted 2024-04-10 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenofovir (Experimental): patients with parkinson's disease
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- Placebo (Placebo Comparator): patients with parkinson's disease
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — take tenofovir disoproxil fumarate 300mg/d

SUMMARY:
To evaluate the efficacy and safety of tenofovir disoproxil fumarate in the treatment of Parkinson's disease. The changes of motor symptoms and the occurrence of adverse reactions in early Parkinson's disease patients who took tenofovir disoproxil fumarate and did not take Tenofovir disoproxil fumarate at different time points were compared.

ELIGIBILITY:
Inclusion Criteria:

* 1: Parkinson's disease: Hoehn Yahr= 1 to 2.5 2: MMSE score≥24

Exclusion Criteria:

* 1: essential tremor, stroke, epilepsy and other well-defined neurological disorders

  2: Or have received deep brain stimulation and other brain surgery

  3: Abnormal liver and kidney function

  4: Infected with chronic hepatitis B or AIDS (HIV-1 infection)

  5: Severe depression, schizophrenia, other psychiatric disorders or drug dependence

  6: Other serious physical diseases such as heart, lung, liver, kidney disease, blood disease and malignant tumor

  7: Pregnant or lactating women and seniors over 65 years of age

  8: Allergy or other contraindications to the investigational drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
UPDRS III（Unified Parkinson's Disease Rating Scale part 3） | 1 month、3 month
  score：0-132，higher scores mean a worse outcome

SECONDARY OUTCOMES:
Non-Motor Symptom Scale（NMSS） | 1 month、3 month
  score：0-360，higher scores mean a worse outcome
creatinine(μmoI/L) | 1 month、3 month
  blood biochemistry test，normal<97μmoI/L

CONTACTS AND LOCATIONS:
Locations (1):
- Guohua Zhao, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No